CLINICAL TRIAL: NCT02516228
Title: Geodesic Transcranial Electrical Neuromodulation(GTEN100) Device
Brief Title: Transcranial Electrical Neuromodulation for Suppressing Epileptiform Discharges
Acronym: GTEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to discontinue development of this investigational device
Sponsor: Electrical Geodesics, Inc. (Industry)
Collaborators: Harborview Injury Prevention and Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGI-001
Record Dates: First submitted 2015-07-23; First posted 2015-08-05 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GTEN 100 (Experimental): All patients will receive treatment according to the protocol with the GTEN 100 device, pulsed only.
  Interventions: Device: GTEN 100

INTERVENTIONS:
Device: GTEN 100 — Stimulation will be focused on the seizure generating cortex. All patients enrolled in the study will have a pre-treatment baseline evaluation period. During this time, the patient (and/or family) will maintain the seizure diary that simply tracks the number of seizure the patient experiences each day.
  During this baseline period, two two-hour EEG recordings (to be completed on 2 separate days) will be acquired. This baseline EEG data will be used to establish baseline inter-ictal spike rate as well as classification of the inter-ictal spikes used to localize seizure onset zone. Using the localization information, patients will be treated with the device for five concurrent days.
  Other Names: GTEN

SUMMARY:
This study examines the safety and feasibility of suppressing epileptic discharges through inducing long term depression of the epileptic focus with transcranial electrical neuromodulation.

DETAILED DESCRIPTION:
One third of patients with epilepsy continue to have seizures despite receiving antiepileptic medication. The application of low frequency repetitive transcranial magnetic stimulation (rTMS) has shown promise for decreasing the frequency of epileptic seizures in drug refractory patients. The mechanism of action appears to be induction of long term depression (LTD) in the targeted cortex by the low frequency (0.5 Hz or 1 every 2 sec) pulses. Unfortunately, the electrical stimulation induced by available TMS coils is limited to the most superficial (gyral) regions of cortex, whereas epileptic foci may occur in sulci, and in deep as well as superficial cortex. The investigators have developed the ability to target currents to specific regions of cortex by aligning source and sink electrodes with flexible subsets of a 256 channel geodesic electrode array. A first step is accurate localization of the likely epileptic focus with 256 channel EEG. Detailed computational models of the electrical properties of head tissues allow optimization studies to select the best pattern of source-sink electrodes for that individual's head tissues and epileptic focus. The goal of the safety and feasibility trial is to test whether one week (5 days) of GTEN treatment can achieve a similar depression of the target cortical region as low frequency rTMS, with the decrease in excitability measured by suppression of epileptic spikes. This safety and feasibility trial has received an Investigational Device Exemption from the FDA for treating 20 patients with focal neocortical epilepsy. Pulsed (emulating rTMS) current sequences will be evaluated. The GTEN system implements a number of advanced technologies that provide improved targeting compared to conventional rTMS or tDCS, including electronics for both pulsed and sustained delivery of current with 256 electrodes; double fault safety circuits; computational modeling of the electromagnetic properties of the patient's head tissue for GTEN targeting with medical grade software; a lidocaine electrolyte that minimizes pain of the pulsed or sustained current with up to 200 µA per electrode (2 mA total); and online safety monitoring for adverse EEG changes with the 256 dEEG array. Based on FDA feedback to date, success with these trials will allow us to progress to a pivotal clinical efficacy trial (with separate funding) to support a de novo 510k approval for GTEN treatment for the temporary suppression of seizures in patients with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14 to 60.
2. Partial onset seizures (simple or complex) with failure of adequate seizure control after prior use of at least 2 anti-seizure drugs at effective doses.
3. Only one clearly identified and localizable extratemporal focus of epileptiform discharges, as defined the discharges (typically epileptiform spikes) and as identified by dEEG assessment through one or more routine clinical dEEG evaluations.
4. Two or more partial seizures, with or without secondary generalization, in the last month, but less than 10 seizures per day.
5. Anti-seizure drug regimen has remained unchanged for the month before study entry, and there is reasonable likelihood of stability for the duration of the study, with the exception of allowing short-term rescue medications, such as lorazepam.
6. A history of epilepsy for at least 2 years.

Exclusion Criteria:

1. Patient is pregnant or becomes pregnant
2. A history or condition of progressive brain disorders, unstable systemic diseases, symptomatic cerebrovascular disease, cardiac disease, or alcohol/substance abuse.Special conditions, for example, non-malignant brain tumors and vascular malformations, can be considered for entry on a case-by-case basis.
3. A history or condition of status epilepticus or psychogenic seizures (seizures not confirmed by EEG).
4. Presence of a cardiac pacemaker, vagus nerve stimulator, or metal implants in the body (other than the teeth) including neurostimulators, cochlear implants, and implanted medication pumps (screened using the LCNI Safety Screening Questionaire).
5. Previous surgery involving opening the skull.
6. Allergy to or condition contraindicating lidocaine.
7. Unable to express presence of pain or discomfort.
8. Allergy to silver
9. Participating in other competing clinical trials
10. Unable to speak English
11. Unable to knowingly give consent

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don M Tucker, Ph.D, Principal Investigator — C.E.O/, Chief Scientist
Locations (1):
- Harborview Medical Center - University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and treatment procedures were conducted in the Neurology clinic at Harborview Hospital. Six subjects were screened and enrolled from 12-02-15 to 04-28-17.
Groups:
- GTEN 100: All patients will receive treatment according to the protocol with the GTEN 100 device, pulsed only.
  GTEN 100: Stimulation will be focused on the seizure generating cortex. All patients enrolled in the study will have a pre-treatment baseline evaluation period. During this time, the patient (and/or family) will maintain the seizure diary that simply tracks the number of seizure the patient experiences each day.
  During this baseline period, two two-hour EEG recordings (to be completed on 2 separate days) will be acquired. This baseline EEG data will be used to establish baseline inter-ictal spike rate as well as classification of the inter-ictal spikes used to localize seizure onset zone. Using the localization information, patients will be treated with the device for five concurrent days.
Period: Overall Study
Arm/Group | GTEN 100
Started | 6
Completed | 3
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | GTEN 100
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 39.3 [22 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Temporary suppression of epileptic spikes [Mean (Standard Deviation); unit: spikes per hour] — Population: This study was running at the time of acquisition by Philips. The study execution was out of compliance from the regulations and GCP. There was no protocol, no statistical analysis plan, no case report forms and no data was formally collected therefore, no statistical analysis was performed. Philips terminated the study.

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Spikes Per Hour
Description: The main efficacy endpoint will be the change from baseline in number of spikes per hour (spike rate), as assessed with routine dEEG sessions, at each visit and after each treatment sessions.
Time Frame: Baseline and following the 5 day treatment session
Population: This study was running at the time of acquisition by Philips. The study execution was out of compliance from GCP. There was no protocol, no statistical analysis plan, no case report forms and no data was collected therefore, no statistical analysis was performed. Philips terminated the study.
Arm/Group | GTEN 100
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Seizures
Description: Weekly change in the number of seizures, assessed by the seizure diary in comparison to the mean weekly seizure frequency for the baseline evaluation period;
Time Frame: Baseline measurement and the Nine Month visit
Population: This study was running at the time of acquisition by Philips. The study execution was out of compliance from the regulations and GCP. There was no protocol, no statistical analysis plan, no case report forms and no data was collected therefore, no statistical analysis was performed. Philips terminated the study.
Arm/Group | GTEN 100
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Cognitive Function Test Score
Description: Change of cognitive function testing score beyond the practice effect (estimated from norms) ;
Time Frame: Nine months
Population: This study was running at the time of acquisition by Philips. The study execution was out of compliance from the regulations and GCP. There was no protocol, no statistical analysis plan, no case report forms and no data was monitored or collected therefore, no statistical analysis was performed. Philips terminated the study.
Arm/Group | GTEN 100
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Quality of Life Rating
Description: Change from baseline in quality of life rating
Time Frame: Nine months
Population: as for outcome 3
Arm/Group | GTEN 100
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Spike Count Suppression
Description: • With assessments of spike rates after treatment session and at visits at weeks 2, 4, 8, 16, and 24, the duration of any suppression in spike rate can be explored. All spike rates (baseline, treatment, and follow-up) will also be classified in relation to waking or sleep stage (N1, N2, N3).
Time Frame: Measured at baseline. treatment and at the 9 month followup visit
Population: as for outcome 3
Arm/Group | GTEN 100
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | GTEN 100
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GTEN 100 (N=6)
Seizure (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02516228/ICF_000.pdf
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT02516228/Prot_001.pdf